CLINICAL TRIAL: NCT05831527
Title: An Exploratory Investigation of a Supplement to Promote Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armra (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20255
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Symptoms; Exercise Performance

STUDY DESIGN:
Intervention Model Description: Multiarm study, both arms receiving the same intervention drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gut Health Group (Experimental): Subjects with self-reported digestive issues (abdominal pain, gas production, bloating after meals, or heartburn after meals) Dose: two sachets daily (1g each) mixed with a cold drink, for 12 weeks.
  Interventions: Drug: ARMRA™ Bovine Colostrum
- Exercise Performance Group (Experimental): Subjects that are physically active three or more days a week. Dose: two sachets daily (1g each) mixed with a cold drink, for 12 weeks.
  Interventions: Drug: ARMRA™ Bovine Colostrum

INTERVENTIONS:
Drug: ARMRA™ Bovine Colostrum — Participants have the option to choose between unflavoured ARMRA™ Bovine Colostrum or blood orange flavoured ARMRA™ Bovine Colostrum.
  Participants took 2 sachets (1g each) of the product mixed with a cold drink daily for 12 weeks.

SUMMARY:
Bovine colostrum is a dairy food and the first milk produced by the mother cow. Abundant research exists revealing the valuable health benefits it confers due to its unique nutritional properties., including benefits to gastrointestinal health, fitness, and overall well-being.This study aims to test a specific food-grade supplement, ARMRA Colostrum Immune Revival, over a 12-week trial to better understand the well-being, fitness, and gut benefits. This trial will use two groups, one that suffers from gastrointestinal complaints frequently and another that exercises at least three days a week.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 18-65 years of age.
* Self-reported digestive issues (abdominal pain, gas production, bloating after meals, or heartburn after meals) (GUT HEALTH GROUP ONLY)
* Must be physically active three or more days a week and willing to maintain their current activity level (PERFORMANCE GROUP ONLY)
* Must be willing to refrain from lifestyle changes affecting their gastrointestinal tract.
* Must be in good health with no significant chronic conditions.
* Following a stable, consistent diet regimen.
* Have a reliable way to measure their weight.

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Suffers from pre-existing conditions that would prevent them from adhering to the protocol.
* Has a lactose allergy or intolerance.
* Serious food allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Change in overall well-being [Time Frame: Baseline to Week 12] | 12 weeks
  Well-being will be measured via study-specific surveys. Data was collected using a textual 5 or 6-point Likert scale for each question, such as "Not noticeable" to "severe." Symptom-related questions were conducted at baseline and each check-in. The textual Likert data was transformed into numerical values of 1-6, with 1 representing the least favorable/worse outcome ("severe" response to the question, "how severe would you rate your stress"), and 6 representing the most beneficial response (i.e., "no symptoms" to the question, "how severe would you rate your stress").
Change in hs-CRP [Time Frame: Baseline to Week 12] | 12 weeks
  Biomarker assessment will be completed to assess changes in hs-CRP. Participants will complete a finger-prick dried blood spot test, at Baseline and Week 12.

SECONDARY OUTCOMES:
Change in self-reported gastrointestinal outcomes, such as bloating, heartburn, irregular bowel movements, and gas [Time Frame: Baseline to Week 12] | 12 weeks
  In the Gut Health Group only: Assessed via self-reported gastrointestinal outcomes such as bloating, heartburn, irregular bowel movements, and gas. Data was collected using a textual 5 or 6-point Likert scale for each question, such as "Not noticeable" to "severe." Symptom-related questions were conducted at baseline and each check-in. The textual Likert data was transformed into numerical values of 1-6, with 1 representing the least favorable/worse outcome ("severe" response to the question, "how severe would you rate your stress"), and 6 representing the most beneficial response (i.e., "no symptoms" to the question, "how severe would you rate your stress").
Change in recovery and fitness levels [Time Frame: Baseline to Week 12] | 12 weeks
  In the Exercise Performance Group only: Assessed via self-reported questionnaires. Data was collected using a textual 5 or 6-point Likert scale for each question, such as "Not noticeable" to "severe." Symptom-related questions were conducted at baseline and each check-in. The textual Likert data was transformed into numerical values of 1-6, with 1 representing the least favorable/worse outcome ("severe" response to the question, "how severe would you rate your stress"), and 6 representing the most beneficial response (i.e., "no symptoms" to the question, "how severe would you rate your stress").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States